CLINICAL TRIAL: NCT05781256
Title: Study on the Association Between Sleep Blood Pressure Patterns and Blood Pressure Values in Daily Life - Usefulness of Novel BP Monitoring Methods
Brief Title: Novel BP Monitoring Methods to Study the Association Between Sleep BP Patterns and BP Values in Daily Life
Acronym: CABER-NET
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09J902
Record Dates: First submitted 2022-06-16; First posted 2023-03-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Ambulatory Blood Pressure Monitoring; Home Blood Pressure Monitoring; Blood Pressure Determination; Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Out-of-office blood pressure (BP) measurement by means of ambulatory BP monitoring (ABPM) or home BP monitoring (HBPM) is recommended for the diagnosis and management of hypertension in the latest guidelines. Ambulatory BP values are more strongly associated with target organ damage and cardiovascular (CVD) events than office values. In particular, nocturnal blood pressure level and reduction of BP during the night (dipping) have been recognised as predictors of cardiovascular complications. However, in current clinical practice, these parameters are derived from ABPM. HBPM represents an inexpensive alternative to ABPM, is preferred by patients and provides a more realistic assessment of BP during an individual's daily life. However, until recently, HBPM did not offer the possibility to measure nocturnal BP or dipping.

The development and validation of new BP devices, such as the NightView (OMRON Healthcare, HEM9601T-E3) could overcome this limitation, offering the possibility of home night-time BP measurements with minimal sleep disturbance. On the other hand the use of wearable devices such as HeartGuide (OMRON Healthcare, HEM-6411T-MAE) could provide BP values in daily life conditions. Compared with conventional HBP, typically measured in resting conditions at home, values obtained with wearable devices might be closer to daytime ABP values.

Combining nocturnal HBP, with daytime BP from wearable device could therefore allow the estimation of dipping status comparable with that provided by ABPM.

In order to compare HBP-derived dipping estimate with the gold standard ABPM-derived value, it is aimed to enrol patients with hypertension, assess their blood pressure profile with ABPM and provide them with both NightView and HeartGuide devices for 7 days. Then diurnal and nocturnal BP and dipping derived from standard 24-hour ABPM will be compared and the combination of NightView/HeartGuide in order to understand whether the latter can offer a reliable assessment of 24h BP pattern.

For a better phenotypization of nocturnal BP and dipping status the following determinants of nocturnal BP and dipping status will be also investigated: sleep quality, sleep duration, the presence of sleep disorders, salt consumption, catecholamine phenotype.

This study will offer the unique opportunity to understand whether such new HBP devices can be offered in alternative to ABPM in the assessment of 24h BP profile in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* arterial hypertension defined as office systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg or the presence of antihypertensive treatment
* antihypertensive treatment stable over 2 weeks preceding enrolment
* written informed consent

Exclusion Criteria:

* atrial fibrillation/flutter of frequent ectopic beats
* pregnancy and lactation
* terminal malignant disease, life expectancy <6 months
* limb amputation
* dementia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * >18 years old
  * arterial hypertension defined as office systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg or the presence of antihypertensive treatment
  * antihypertensive treatment stable over 2 weeks preceding enrolment
  * written informed consent
  Exclusion Criteria:
  * atrial fibrillation/flutter of frequent ectopic beats
  * pregnancy and lactation
  * terminal malignant disease, life expectancy <6 months
  * limb amputation
  * dementia
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Nocturnal blood pressure fall - wearable validated device | 1 week
  Average nocturnal blood pressure fall, assessed through a validated wearable device over 7 days
Nocturnal blood pressure fall - ABPM | 1 week
  Average nocturnal blood pressure fall, assessed through ABPM over 7 days

SECONDARY OUTCOMES:
Average sleep duration | 1 week
  Average sleep duration in hours over 7 days, measured by simplified polysomnography
Average systolic and diastolic blood pressure - wearable validated device | 1 week
  Average systolic and diastolic blood pressure in daily life conditions, assessed through a validated wearable device over 7 days
Average systolic and diastolic blood pressure - ABPM | 1 week
  Average systolic and diastolic blood pressure in daily life conditions, assessed through ABPM over 7 days
Leptin levels | At baseline
  Leptin levels at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martino Pengo, MD, PhD, Study Chair — Istituto Auxologico Italiano
Locations (1):
- Martino Pengo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No